CLINICAL TRIAL: NCT06458738
Title: Clinical Evaluation of a New Printable Denture Base Material: a Prospective Single-arm Study
Brief Title: Clinical Evaluation of a New Printable Denture Base Material
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTCS 11891315
Record Dates: First submitted 2024-06-06; First posted 2024-06-14 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Printable denture base material (Experimental)
  Interventions: Device: Printable denture base material

INTERVENTIONS:
Device: Printable denture base material — The newly developed printable denture base material will be used for the production of dentures.

SUMMARY:
This clinical investigation is conducted to prove the long-term clinical performance of a new printable denture base material. The aim of this study is to assess the failure rate, the quality and functionality of the full dentures made with the printable denture base material over an investigational period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 84 years
* informed consent signed and understood by the subject
* full edentulous patients
* a digital design of the dentures is already existing.
* ability to visit the clinic in person until the baseline recall

Exclusion Criteria:

* patient does not wear the dentures regularly
* mental health status does not allow reliable feedback
* patients with a proven allergy to one of the ingredients (methacrylates) of the materials used
* patients with severe systemic diseases
* poor oral / denture hygiene
* pregnancy

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
rate of failures leading to replacement of denture | 5 years
  number of dentures

SECONDARY OUTCOMES:
functional (e.g. retention) properties of the dentures | 5 years
  Evaluated according to adapted FDI criteria (grade 1-4). Lower scores mean a better outcome.
biological (e.g. plaque accumulation) properties of the dentures | 5 years
  Evaluated according to adapted FDI criteria (grade 1-4). Lower scores mean a better outcome.
aesthetic (e.g. surface staining) properties of the dentures | 5 years
  Evaluated according to adapted FDI criteria (grade 1-4). Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent AG, Schaan, Liechtenstein, Liechtenstein

IPD SHARING:
Plan to Share IPD: No